CLINICAL TRIAL: NCT01577745
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI0639 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI0639 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI0639-1078
Record Dates: First submitted 2012-04-05; First posted 2012-04-16 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Solid Tumors
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MEDI0639 Cohort 1 (Experimental): Participants received MEDI0639 dose level 1 as a 60-minute intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: MEDI0639
- MEDI0639 Cohort 2 (Experimental): Participants received MEDI0639 dose level 2 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: MEDI0639
- MEDI0639 Cohort 3 (Experimental): Participants received MEDI0639 dose level 3 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: MEDI0639
- MEDI0639 Cohort 4 (Experimental): Participants received MEDI0639 dose level 4 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: MEDI0639
- MEDI0639 Cohort 5 (Experimental): Participants received MEDI0639 dose level 5 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: MEDI0639
- MEDI0639 Cohort 6 (Experimental): Participants received MEDI0639 dose level 6 as a 60-minute IV infusion on Day 1 of each 21 day cycle.
  Interventions: Biological: MEDI0639

INTERVENTIONS:
Biological: MEDI0639 — MEDI0639 is an immunoglobulin G1 lambda (IgG1λ) monoclonal antibody. MEDI0639 selectively binds to DLL4 and blocks its ability to bind to and activate signaling through the Notch receptors.

SUMMARY:
This is a first-time-in-human, Phase 1, multicenter, open-label, single-arm, dose-escalation (3+3) study to evaluate the safety, tolerability, antitumor activity, PK and immunogenicity of MEDI0639.

DETAILED DESCRIPTION:
This is a first-time-in-human, Phase 1, multicenter, open-label, single-arm, dose-escalation (3+3) study to evaluate the safety, tolerability, antitumor activity, PK, and immunogenicity of MEDI0639 in adult subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy exist. Up to 63 subjects will be enrolled at approximately 3 to 5 study centers in North America.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors that are refractory to standard therapy or for which no standard therapy exist
* Age ≥ 18 years
* ECOG Performance Status of 0 or 1
* LVEF (measured by Echocardiogram) > 50%
* No gastrointestinal bleeding within 1 year of study entry.
* Adequate organ and marrow function:

  * Hemoglobin ≥ 10g/dL
  * Absolute Neutrophil Count ≥ 1500/mm3
  * Platelet Count ≥ 100,000/mm3
  * AST & ALT ≤ 2.5 x ULN
  * Bilirubin ≤ 1.5 x ULN
  * Cr Cl ≥ 50 mL/min (as determined by the Cockcroft-Gault equation or by 24-hour urine collection)
* Prior therapy against VEGF or VEGFRs including, but not limited to bevacizumab, sunitinib, sorafenib, pazopanib, motesanib (AMG706), or cediranib (AZD2171), is permitted so long as the agent does not have any known activity against DLL4 and the last dose received s at least 6 weeks prior to first dose of MEDI0639.
* Life expectancy ≥ 12 weeks
* Females of childbearing potential must be surgically sterile, have a sterile male partner, be premenarchal or at least 2 years postmenopausal, practice abstinence or otherwise must use 2 effective methods of contraception from the time of initiation of investigational product.
* Males, unless surgically sterile, must use 2 effective methods of contraception with a female partner and must agree to continue using such contraception for 90 days after the last dose of MEDI0639

Exclusion Criteria:

* Concurrent enrollment in another investigational clinical study
* Receipt of any investigational anticancer therapy within 4 weeks prior to the first dose of MEDI0639 or in the case of monoclonal antibodies, 6 weeks prior to the first dose of MEDI0639
* Concurrent or previous treatment with inhibitors of DLL4
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment
* Known bleeding diathesis, esophageal varices, or angioplasty
* Pulmonary hemorrhage or gross hemoptysis within 12 months
* Known arterial or venous thrombosis or pulmonary embolism within 2 years
* Concurrent use of systemic low molecular weight heparin or low dose warfarin
* Presence of brain metastases
* Cerebrovascular accident or transient ischemic attack within 2 years
* Cardiovascular events, such as myocardial infarction, unstable/severe angina, coronary/peripheral artery bypass graft, unstable cardiac arrhythmia requiring medication, congestive heart failure (NYHA > class II), within 2 years
* Tumors with squamous cell histology
* Major surgical procedure within 90 days
* Pregnancy or lactation
* Known HIV positive or Hepatitis A, B, or C infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 58 participants were screened at 7 sites in the United States of America (USA).
Pre-assignment Details: A total of 58 participants were screened for this study, of which 25 participants were enrolled and received study treatment.
Period: Overall Study
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Started | 3 | 3 | 3 | 6 | 5 | 5
Completed | 0 | 0 | 1 | 0 | 0 | 1
Not Completed | 3 | 3 | 2 | 6 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 3 | 2 | 0
Not completed — Death | 3 | 2 | 2 | 1 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Alternative Therapy | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of MEDI0639.
Groups:
- MEDI0639 Cohort 1: Participants received MEDI0639 dose level 1 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (14.0) | 57.3 (22.5) | 67.7 (13.7) | 62.2 (9.3) | 62.2 (5.2) | 62.6 (10.8) | 61.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 3 | 3 | 3 | 13
  Male | 3 | 0 | 2 | 3 | 2 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 2 | 3 | 6 | 4 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 3 | 2 | 3 | 6 | 5 | 5 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MEDI0639
Description: The MTD evaluation was based on the dose-limiting toxicity (DLT) evaluable population. DLT is defined as any Grade 3 or higher treatment-related toxicity that occurred during the DLT evaluation period (defined as the time from the first dose of MEDI0639 to 21 days after the first dose), except for National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 hypertension that could be controlled within 96 hours; Grade 3 symptomatic hypertension of greater than (>) 180 millimetre of mercury (mm Hg) systolic or >120 mm Hg diastolic or asymptomatic hypertension of >200 mm Hg systolic or >120 mm Hg diastolic was considered a DLT.
Time Frame: From the first dose of MEDI0639 to 21 days after the first dose
Population: All participants enrolled in the dose-escalation phase who received at least 1 full cycle of MEDI0639 and completed safety follow-up through the DLT evaluation period or experienced any DLT.
Measure: Number; unit: milligram (mg)
Groups:
- MEDI0639: Participants received MEDI0639, in dose escalation phase starting from dose level 1 to 6 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
Arm/Group | MEDI0639
Number analyzed (Participants) | 25
milligram (mg) | NA — There were no participants with DLTs, hence MTD was not identified. The maximum administered dose was 200 mg.

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug. Treatment-emergent AEs (TEAEs) were events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, for the period extending to 90 days after the last dose of study drug. The AEs were summarized using Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.
Time Frame: From the first dose of MEDI0639 until 90 days after the last dose of MEDI0639. Maximum time frame across participants was 11 months.
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
participants | 3 | 3 | 3 | 6 | 5 | 5

3. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: A serious AE (SAE) is any AE that results in death (refers to an event, which risk of death at the time of the event; it does not refer to an event that may have led to death), is immediately life threatening, require (or prolong) inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above. Treatment-emergent SAEs defined as SAEs present at baseline that worsened in intensity after administration of study drug or SAEs absent at baseline that emerged after administration of study drug. The SAEs were summarized using MedDRA version 18.1.
Time Frame: From the first dose of MEDI0639 until the end of participation in the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Participants
Groups:
- MEDI0639 Cohort 6: Participants received MEDI0639 dose level 6 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants | 2 | 1 | 2 | 2 | 4 | 3

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Laboratory Parameters
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (white blood cell [WBC] count with differential, red blood cell [RBC] count, hematocrit, hemoglobin, platelet count, mean corpuscular volume [MCV], and mean corpuscular hemoglobin concentration [MCHC]); serum chemistry (calcium, chloride, magnesium, potassium, sodium, bicarbonate, aspartate transaminase [AST], alanine transaminase [ALT], alkaline phosphatase, total bilirubin, liver function test, gamma glutamyl transferase [GGT], lactate dehydrogenase, uric acid, creatinine, blood urea nitrogen [BUN], glucose, albumin, total protein, triglycerides, cholesterol, and troponin); and routine urinalysis. The TEAEs related to laboratory evaluations in participants were reported.
Time Frame: From the first dose of MEDI0639 until 90 days after last dose of MEDI0639. Maximum time frame across participants was 11 months.
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants
  Anaemia | 2 | 0 | 0 | 3 | 3 | 1
  Leukocytosis | 1 | 1 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 0 | 1 | 0
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 2
  Neutropenia | 0 | 0 | 0 | 0 | 1 | 0
  Thrombocytopenia | 0 | 1 | 0 | 0 | 1 | 0
  White blood cell count decreased | 0 | 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase increased | 0 | 1 | 2 | 0 | 0 | 1
  Aspartate aminotransferase increased | 1 | 2 | 2 | 1 | 0 | 2
  Blood alkaline phosphatase increased | 1 | 0 | 2 | 2 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0
  Blood cholesterol increased | 0 | 0 | 1 | 0 | 0 | 0
  Blood creatinine increased | 0 | 0 | 0 | 1 | 0 | 0
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 1
  Blood triglycerides increased | 1 | 0 | 1 | 0 | 0 | 0
  Brain natriuretic peptide increased | 1 | 1 | 0 | 2 | 2 | 0
  Gamma-glutamyltransferase increased | 3 | 1 | 2 | 2 | 0 | 0
  N-terminal prohormone BNP increased | 0 | 0 | 1 | 0 | 0 | 0
  Troponin I increased | 2 | 0 | 0 | 0 | 0 | 0
  Troponin increased | 0 | 0 | 0 | 0 | 0 | 1
  Hepatobiliary disorders | 1 | 0 | 0 | 0 | 1 | 0
  Hyperbilirubinaemia | 1 | 0 | 0 | 0 | 0 | 0
  Metabolism and nutrition disorders | 2 | 3 | 3 | 3 | 3 | 2
  Dyslipidaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypercalcaemia | 0 | 0 | 0 | 1 | 1 | 0
  Hypercholesterolaemia | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0 | 1 | 0
  Hyperkalaemia | 1 | 0 | 1 | 0 | 1 | 0
  Hypernatraemia | 0 | 0 | 1 | 0 | 0 | 0
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypertriglyceridaemia | 0 | 0 | 1 | 0 | 1 | 0
  Hyperuricaemia | 0 | 1 | 1 | 0 | 0 | 0
  Hypoalbuminaemia | 1 | 1 | 0 | 0 | 0 | 1
  Hypocalcaemia | 0 | 0 | 1 | 0 | 0 | 0
  Hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 1
  Hypokalaemia | 0 | 1 | 0 | 0 | 0 | 0
  Hypomagnesaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hyponatraemia | 0 | 1 | 0 | 1 | 0 | 0
  Hypophosphataemia | 0 | 0 | 0 | 1 | 0 | 0
  WBC urine positive | 0 | 0 | 1 | 0 | 0 | 0
  Proteinuria | 1 | 1 | 0 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Vital Signs and Physical Examination
Description: Vital signs (temperature, blood pressure, pulse rate, and respiratory rate) were performed at baseline and throughout the study. The TEAEs related to vital signs in participants were reported.
Time Frame: as for outcome 4
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants
  Electrocardiogram QT prolonged | 1 | 1 | 0 | 2 | 0 | 0
  Weight decreased | 1 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram t wave amplitude decreased | 0 | 1 | 0 | 0 | 0 | 0
  Hypotension | 0 | 1 | 1 | 0 | 0 | 0
  Pyrexia | 0 | 2 | 0 | 2 | 2 | 0
  Atrial fibrillation | 0 | 0 | 1 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 2 | 1 | 1
  Atrioventricular block first degree | 0 | 0 | 0 | 1 | 0 | 0
  Electrocardiogram ST-T change | 0 | 0 | 0 | 1 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Electrocardiogram (ECG) Evaluations
Description: ECG parameters included QT interval and corrected QT (QTc) interval. Electrocardiogram (ECG) parameters were assessed at baseline as well as throughout the study. All 12-lead ECGs performed during the study were obtained in triplicate. The TEAEs related to ECG evaluations in participants were reported.
Time Frame: as for outcome 4
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants
  ECG QT prolonged | 1 | 1 | 0 | 2 | 0 | 0
  Electrocardiogram t wave amplitude decreased | 0 | 1 | 0 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 1 | 0 | 0 | 0
  Atrioventricular block first degree | 0 | 0 | 0 | 1 | 0 | 0
  Electrocardiogram ST-T change | 0 | 0 | 0 | 1 | 0 | 0

7. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Echocardiogram Evaluations
Description: Echocardiogram parameters included left ventricular ejection fraction (LVEF) and pulmonary arterial pressure (PAP). The TEAEs related to echocardiogram evaluations in participants were reported.
Time Frame: as for outcome 4
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) After Cycle 1 Treatment Administration of MEDI0639
Description: The pharmacokinetics (PK) parameter was estimated using the noncompartmental analysis methods, based on the individual serum concentration-time data. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI0639.
Time Frame: Days 1 (prior to start of infusion and 30 mins, 2, and 6 hours post end of infusion), 2, 5 , 8, and 15 of Cycle 1
Population: All the participants who received dose of MEDI0639 in Cycle 1 and for whom Pharmacokinetic (PK) blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter (mcg*d/mL)
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
microgram*day per milliliter (mcg*d/mL) | 7.41 (1.04) | 41.1 (34.0) | 89.9 (64.9) | 179 (59.9) | 434 (91.9) | 512 (250)

9. Secondary Outcome: Maximum Observed Concentration (Cmax) After Cycle 1 Treatment Administration of MEDI0639
Description: as for outcome 8
Time Frame: Days 1 (prior to start of infusion and 30 mins, 2, and 6 hours post end of infusion), 2, 5 , 8, and 15 of Cycle 1
Population: All the participants who received dose of MEDI0639 in Cycle 1 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
microgram per milliliter (mcg/mL) | 3.19 (0.759) | 11.8 (2.45) | 18.3 (4.96) | 27.2 (7.32) | 60.5 (13.5) | 81.6 (47.3)

10. Secondary Outcome: Clearance (CL) After Cycle 1 Treatment Administration of MEDI0639
Description: The pharmacokinetics (PK) parameter was estimated using the noncompartmental analysis methods, based on the individual serum concentration-time data. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI0639. Clearance was estimated as dose divided by the area under serum concentration-time curve from time zero to infinity.
Time Frame: Days 1 (prior to start of infusion and 30 mins, 2, and 6 hours post end of infusion), 2, 5 , 8, and 15 of Cycle 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liter per day (L/d)
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Liter per day (L/d) | 1.37 (0.182) | 1.06 (0.602) | 0.895 (0.480) | 0.619 (0.230) | 0.360 (0.0860) | 0.504 (0.330)

11. Secondary Outcome: Half-life (t1/2) After Cycle 1 Treatment Administration of MEDI0639
Description: as for outcome 8
Time Frame: Days 1 (prior to start of infusion and 30 mins, 2, and 6 hours post end of infusion), 2, 5 , 8, and 15 of Cycle 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Days | 1.50 (0.193) | 2.53 (0.580) | 5.09 (3.43) | 6.42 (1.93) | 9.74 (2.26) | 8.25 (3.11)

12. Secondary Outcome: Number of Participants Positive With Antidrug Antibodies (ADA) for MEDI0639
Description: Blood samples were measured for the presence of ADA for MEDI0639 using a validated bridging immunoassay. Only the number of participants positive for anti-MEDI-575 antibodies at any visit were presented.
Time Frame: On Day 1 of Cycles 1, 2, 3, and every other cycle thereafter, end of treatment, 30 days, and 3 and 6 months after the last dose of MEDI0639. Maximum time frame across participants was 14 months.
Population: All participants who received any treatment with MEDI0639.
Measure: Number; unit: Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Percentage (%) of participants who were responders with BOR documented as confirmed CR, PR, stable disease (SD), progressive disease (PD) and non-evaluable (NE). CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. PR: At least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Percentage of Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 33.3 | 0 | 0 | 0
  Stable Disease (SD) | 66.7 | 33.3 | 33.3 | 33.3 | 80.0 | 0
  Progressive Disease (PD) | 33.3 | 66.7 | 33.3 | 66.7 | 20.0 | 60.0
  Non-Evaluable (NE) | 0 | 0 | 0 | 0 | 0 | 40.0

14. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate (ORR) defined as the percentage of participants with a BOR of confirmed CR or confirmed PR.
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639. All participants with an objective response were included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- MMEDI0639 Cohort 5: Participants received MEDI0639 dose level 5 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
- MMEDI0639 Cohort 6: Participants received MEDI0639 dose level 6 as a 60-minute IV infusion on Day 1 of each 21-day cycle.
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MMEDI0639 Cohort 5 | MMEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Percentage of Participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2]

15. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control rate (DCR) defined as the percentage of participants with a BOR of confirmed CR, confirmed PR or SD.
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Percentage of Participants | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 33.3 [4.3 to 77.7] | 80.0 [28.4 to 99.5] | 0 [0.0 to 52.2]

16. Secondary Outcome: Time to Response
Description: Time to response (TTR) defined as the time from the first dose of MEDI0639 until the first documentation of a subsequently confirmed objective response. Only participants who have achieved objective response (confirmed CR or confirmed PR) was evaluated for TTR. TTR (months) = (Date of first disease response - Date of the first dose of MEDI0639 + 1) / (365.25/12).
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639. All participants with an objective response were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
Months |  |  | 1.3 [NA to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint |  |  |

17. Secondary Outcome: Duration of Response (DR)
Description: DR defined as time from start of first documented objective response [confirmed Complete Response (CR) or confirmed Partial Response (PR)] to first documented disease progression or death due to any cause, whichever occurs first. DR calculated as (months) = (Date of PD/death or censoring - Date of first disease response + 1)/ (365.25/12).
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639. All participants with an objective response were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
Months |  |  | 5.9 [NA to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint |  |  |

18. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the first dose of MEDI0639 until the first documentation of disease progression or death due to any cause, whichever occurs first. PFS (months) = (Date of PD/death or censoring - Date of the first dose of MEDI0639 + 1) / (365.25/12).
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Months | 5.1 [1.2 to 5.1] | 1.3 [1.3 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | 7.1 [1.3 to 7.2] | 1.3 [0.7 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | 4.8 [1.4 to 4.8] | 0.9 [0.7 to 1.4]

19. Secondary Outcome: Overall Survival
Description: Overall survival defined as the time from the first dose of MEDI0639 until death due to any cause. OS (months) = (Date of death or censoring - Date of the first dose of MEDI0639 + 1) / (365.25/12).
Time Frame: From study entry through the end of the study. Maximum time frame across participants was 4 years.
Population: All participants who received at least one dose of MEDI0639.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 5 | 5
Months | 6.1 [5.1 to 7.2] | NA [7.8 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | 28.9 [13.8 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | NA [3.5 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | 19.9 [NA to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint | 3.0 [1.1 to NA] — Not evaluable due to insufficient numbers of participants achieved endpoint

ADVERSE EVENTS:
Time Frame: AEs collected from first dose of MEDI0639 to 90 days post dose of MEDI0639, max time frame across participants was 11 months. SAEs collected from the first dose of MEDI0639 to end of participation in study; max time frame across participants was 4 yrs.
Arm/Group | MEDI0639 Cohort 1 | MEDI0639 Cohort 2 | MEDI0639 Cohort 3 | MEDI0639 Cohort 4 | MEDI0639 Cohort 5 | MEDI0639 Cohort 6
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 2/6 | 4/5 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0639 Cohort 1 (N=3) | MEDI0639 Cohort 2 (N=3) | MEDI0639 Cohort 3 (N=3) | MEDI0639 Cohort 4 (N=6) | MEDI0639 Cohort 5 (N=5) | MEDI0639 Cohort 6 (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dilatation ventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis pseudomonas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0639 Cohort 1 (N=3) | MEDI0639 Cohort 2 (N=3) | MEDI0639 Cohort 3 (N=3) | MEDI0639 Cohort 4 (N=6) | MEDI0639 Cohort 5 (N=5) | MEDI0639 Cohort 6 (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 3 (4) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 1 (1) | 2 (2) | 3 (4) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (4) | 2 (3) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 2 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
OMs relationship modulation of DLL4-Notch signaling pathway in tumor and clinical response analysis was not conducted due to low number of evaluable tumor samples and low response rate. Study was terminated early due to lack of clinical activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.